CLINICAL TRIAL: NCT00908050
Title: Double-blind, Placeboa-controlled, Randomized Clinical Trial of the Safety and Efficacy of Botulinum Toxin (BOTOX) in Bruxism.
Brief Title: Study of the Safety and Efficacy of Botox in Bruxism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Joseph Jankovic, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-22737
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2023-05-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Bruxism
Keywords: bruxism, botulinum toxin, sleep study
MeSH Terms: conditions — Bruxism | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo arm
- botulinum toxin type A (Active Comparator): Active arm
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Patients are injected with botulinum toxin type A (BOTOX) 60 units in each masseter muscle and 35 in each temporalis muscle, bilaterally.
  Other Names: Botulinum toxin type A (Botox)
  Arms: botulinum toxin type A
Drug: Placebo arm — Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether botulinum toxin helps patients with bruxism.

DETAILED DESCRIPTION:
Bruxism represents involuntary movements of the jaw muscles, resulting in tooth grinding and clenching. Generally it occurs during sleep, but occasionally can be present during the day, so called awake bruxism. Bruxism is a common condition, affecting approximately 8% of all people. It is not known what causes bruxism but it may result in tooth damage, jaw pain, headaches, poor quality sleep and may bother your partner's sleep at night due to the tooth grinding noise. There is no generally accepted treatment for bruxism. Mouth guards and several medications have been tried, but they generally did not work or caused side effects.

Botulinum toxin "Botox" is a natural toxin, which weakens the muscles when injected in very small amounts. It is currently approved and used for the treatment of various conditions involving abnormal muscle spasms, such as neck twisting (torticollis), twitching of the face (hemifacial spasm) or eyes (blepharospasm), headaches, muscles stiffness following strokes, and it has also been used cosmetically for wrinkle removal.

Since bruxism is caused by involuntary spasms of the jaw muscles, botulinum toxin has been tried, initial results showing that it is safe and effective. The injections generally take one week to start working and 2 weeks for a full effect, which lasts on average 12-16 weeks, and slowly wear off. The injections are generally repeated every 3-4 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients between the ages of 18 and 80 years old with a diagnosis of bruxism, based on the standard criteria.
* 2. If the subject is a female of childbearing age, she must have had a hysterectomy, tubal ligation, or otherwise be incapable of pregnancy, or have practiced a method of contraception (hormonal contraceptives, spermicidal barrier, intrauterine device, partner sterility) at least one month prior to study entry. Any female of childbearing age will have a urine pregnancy test one week prior to the treatment (visit 2).
* 3. Ability of the patient or guardian to sign and understand informed consent.
* 4. Ability to follow and comply with study directions.

Exclusion Criteria:

* 1. Coexistence of active psychosis, other active psychiatric disease or cognitive impairment.
* 2. Coexistence of serious co-morbid conditions.
* 3. Exposure to any botulinum toxin preparation within the past 6 months.
* 4. Participation in another experimental therapeutic protocol within 30 days.
* 5. Any medical condition in which the administration of botulinum toxin is contraindicated, including myasthenia gravis, amyotrophic lateral sclerosis or other neuromuscular diseases.
* 6. History of dysphagia.
* 7. History of botulism.
* 8. A condition or situation in which the investigators view will confound the ability of the subject to participate in the study.
* 9. Patients or guardian who are unable to understand and sign informed consent.
* 10. Pregnancy
* 11. Patients who do not meet inclusion criteria.
* 12. Patients in whom it is felt that a major portion of overall sleep morbidity is not related to bruxism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Ondo, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-one subjects were recruited but eight were excluded: 3 prior to randomization/PSG (withdrew consent), 5 before randomization/after PSG (3 for lack of bruxism on PSG, 2 for severe obstructive sleep apnea on PSG with an AHI > 30 / hr).
Groups:
- Botulinum Toxin Type A: botulinum toxin type A (BOTOX)
Period: Overall Study
Arm/Group | Placebo | Botulinum Toxin Type A
Started | 10 | 13
Completed | 10 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Thirty-one subjects were recruited, eight were excluded: 3 (withdrew consent), 5 after PSG (3 for lack of bruxism on PSG, 2 severe OSA on PSG with an AHI > 30 / hr). 19 females were randomized. 21 reported some temporal-mandibular pain. 13 randomized to BoNT-A and 10 randomized to placebo & completed.
Groups:
- Placebo: Placebo arm
  We performed a double blind, placebo-controlled parallel trial of BoNT-A (Botox®, Allergan) for bruxism, followed by an open label extension. Patients were recruited from the Baylor College of Medicine (BCM) Movement Disorders Clinic from April 2009 to March 2011.
- Botulinum Toxin Type A: Active arm
  We performed a double blind, placebo-controlled parallel trial of BoNT-A (Botox®, Allergan) for bruxism, followed by an open label extension. Patients were recruited from the Baylor College of Medicine (BCM) Movement Disorders Clinic from April 2009 to March 2011.
- Total: Total of all reporting groups
Arm/Group | Placebo | Botulinum Toxin Type A | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Bruxism Questionnaire Baseline and at Week 4
Description: Baseline assessments included a bruxism questionnaire with a modified quantifiable portion [Lavigne G. with permission]. This is compared to week 4 assessments. The bruxism questionnaire consists of 8 questions. Each question can be scored between 0-3 points for a total possible scoring of 24 points. The minimum score is 0. The maximum score if 24. A score of 3 or less means non-temporomandibular disorder. A score of 4 or more means temporomandibular disorder.
Time Frame: baseline versus week 4
Population: Bruxism questionnaire comparison at Week 4 in placebo versus active treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo arm at baseline
  Baseline assessments included a bruxism questionnaire with a modified quantifiable portion [Lavigne G. with permission].
- Botulinum Toxin Type A at Baseline; Botulinum Toxin Type A at Week 4: Active arm
  Baseline assessments included a bruxism questionnaire with a modified quantifiable portion [Lavigne G. with permission].
- Placebo Arm at Week 4: Baseline assessments included a bruxism questionnaire with a modified quantifiable portion [Lavigne G. with permission].
Arm/Group | Placebo | Botulinum Toxin Type A at Baseline | Placebo Arm at Week 4 | Botulinum Toxin Type A at Week 4
Number analyzed (Participants) | 10 | 13 | 10 | 13
units on a scale | 19.4 (13.2) | 16.1 (4.1) | 24.0 (5.4) | 24.0 (6.9)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A at Baseline; The averaged data calculated from three nights in each recording period for each subject will be submitted to statistical analysis. Descriptive and non-parametric statistics will be used for the secondary end-points; Test type: Superiority or Other; p = 0.0394, Chi-squared

2. Secondary Outcome: Headache Impact Test (HIT-6) Questionnaire Baseline and at Week 4
Description: Baseline assessments included HIT-6 questionnaire. This is compared to week 4 assessments. The Headache Impact Test consists of 6 questions. Each question can be scored between 6 to 13 points for a possible total of 78 points. A total score of 50 or more means the patient has migraines. A score of 49 or less means the patient has headaches, not migraines. The minimum score if 36. The maximum score is 78 points.
Time Frame: Baseline to week 4
Population: HIT-6 questionnaire comparison at Week 4 in placebo versus active treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo arm at baseline
  Baseline assessments included a HIT-6 questionnaire.
- Botulinum Toxin Type A at Baseline; Botulinum Toxin Type A at Week 4: Active arm
  Baseline assessments included a HIT-6 questionnaire.
- Placebo Arm at Week 4: Baseline assessments included a HIT-6 questionnaire.
Arm/Group | Placebo | Botulinum Toxin Type A at Baseline | Placebo Arm at Week 4 | Botulinum Toxin Type A at Week 4
Number analyzed (Participants) | 10 | 13 | 10 | 13
units on a scale | 57.8 (9.0) | 52.1 (10.6) | 59.2 (9.1) | 51.2 (11.4)

3. Secondary Outcome: Clinical Global Impression (CGI)
Description: With this scale the clinical evaluates the patient and gives the patient a single score based off of the evaluation. The score given can be between 1 and 7 where 1 means the patient is normal and 7 means the patient is amongst the most severely ill. The minimum score if 1. The maximum score is 7.
Time Frame: baseline versus week 4
Population: CGI questionnaire comparison at Week 4 in placebo versus active treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo arm at baseline
  Baseline assessments included a CGI questionnaire.
- Botulinum Toxin Type A at Baseline; Botulinum Toxin Type A at Week 4: Active arm
  Baseline assessments included a CGI questionnaire.
- Placebo Arm at Week 4: Baseline assessments included a CGI questionnaire.
Arm/Group | Placebo | Botulinum Toxin Type A at Baseline | Placebo Arm at Week 4 | Botulinum Toxin Type A at Week 4
Number analyzed (Participants) | 10 | 13 | 10 | 13
units on a scale | 3 (0.05) | 4 (0.05) | 3 (0.05) | 2 (0.05)

4. Secondary Outcome: Visual Analog Scale of Change (VAS)-Pain Scale
Description: Visual Analog scale of change (VAS) (0-100) comparing delta of pre-versus post-injection.The VAS allows the patient to report their current level of pain on a scale of 0-100 where a score of 0-4 means no pain, a score of 5-44 means mild pain, a score of 45-74 means moderate pain and a score of 75-100 means severe pain. The minimum score is 0 and the maximum score if 100.
Time Frame: baseline versus week 4
Population: VAS-pain scale questionnaire comparison at Week 4 in placebo versus active treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo arm at baseline
  Baseline assessments included a VAS-bruxism questionnaire.
- Botulinum Toxin Type A at Baseline; Botulinum Toxin Type A at Week 4: Active arm
  Baseline assessments included a VAS-bruxism questionnaire.
- Placebo Arm at Week 4: Baseline assessments included a VAS-bruxism questionnaire.
Arm/Group | Placebo | Botulinum Toxin Type A at Baseline | Placebo Arm at Week 4 | Botulinum Toxin Type A at Week 4
Number analyzed (Participants) | 10 | 13 | 10 | 13
units on a scale | 47.3 (15.5) | 64.5 (17.8) | 45.8 (19.6) | 48.6 (13.6)

5. Secondary Outcome: Visual Analog Scale of Change (VAS)-Pain
Description: The VAS allows the patient to report their current level of pain on a scale of 0-100 where a score of 0-4 means no pain, a score of 5-44 means mild pain, a score of 45-74 means moderate pain and a score of 75-100 means severe pain. The minimum score is 0 and the maximum sore if 100.
Time Frame: Baseline versus week 4
Population: VAS-pain questionnaire comparison at Week 4 in placebo versus active treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo arm at baseline
  Baseline assessments included a VAS-pain questionnaire.
- Botulinum Toxin Type A at Baseline; Botulinum Toxin Type A at Week 4: Active arm
  Baseline assessments included a VAS-pain questionnaire.
- Placebo Arm at Week 4: Baseline assessments included a VAS-pain questionnaire.
Arm/Group | Placebo | Botulinum Toxin Type A at Baseline | Placebo Arm at Week 4 | Botulinum Toxin Type A at Week 4
Number analyzed (Participants) | 10 | 13 | 10 | 13
units on a scale | 47.3 (15.5) | 44.2 (14.3) | 48.6 (13.6) | 65 (19.6)

ADVERSE EVENTS:
Groups:
- Placebo: Placebo arm
  Baseline assessments included a bruxism questionnaire with a modified quantifiable portion [Lavigne G. with permission]. Additional scales included the Headache Impact Test-6 24, total Pittsburgh Sleep Quality Index 25, Epworth Sleepiness Scale 26, and Self-Rated Anxiety Scale. 27 Subjects then underwent a baseline polysomnogram (PSG) and were excluded if no bruxism was identified, using standard criteria.
- Botulinum Toxin Type A: Active arm
  Baseline assessments included a bruxism questionnaire with a modified quantifiable portion [Lavigne G. with permission]. Additional scales included the Headache Impact Test-6 24, total Pittsburgh Sleep Quality Index 25, Epworth Sleepiness Scale 26, and Self-Rated Anxiety Scale. 27 Subjects then underwent a baseline polysomnogram (PSG) and were excluded if no bruxism was identified, using standard criteria.
Arm/Group | Placebo | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 8/10 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Botulinum Toxin Type A (N=13)
temporal-mandibular pain (General disorders) | 8 (8) | 13 (13)
cosmetic change in smile (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No